CLINICAL TRIAL: NCT05312528
Title: Diagnostic Value of Annexin V, sVCAM-1, sICAM-1, Vascular Endothelial Growth Factor, TNF Alpha and Interleukin-6 in Ovarian and Deep Infiltrating Endometriosis, the Changes of These Markers in the Postoperative Period
Brief Title: Evaluation of New Biomarkers in Stage 3 and 4 Endometriosis
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Evrim Ebru Kovalak, Medical Doctor, Obstetrician and Gynecologist, Bagcilar Training and Research Hospital
Other Study IDs: 2018.01.1.01.001
Record Dates: First submitted 2022-02-23; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Stage 3 and 4 endometriosis patients
  Interventions: Procedure: endometriosis surgery
- Control Group: Patients without endometriosis, who required surgery for tubal ligation, benign ovarian cysts or uterine fibroids were included.
  Interventions: Procedure: other benign condition surgeries

INTERVENTIONS:
Procedure: endometriosis surgery — Laparoscopy was performed in the follicular phase of the woman's menstrual cycle and all recognizable endometriotic lesions were treated by bipolar coagulation, resection of endometriotic nodules and ovarian cystectomy.
  Groups: Study Group
Procedure: other benign condition surgeries — ovarian cystectomy, bilateral tubal ligation, myomectomy etc.
  Groups: Control Group

SUMMARY:
The diagnostic value of Annexin V, sVCAM-1, sICAM-1, vascular endothelial growth factor and Proinflammatory cytokines (TNF-a and interleukin-6) in ovarian endometriosis and deep infiltrating endometriosis, their levels in organ-specific involvement, their relationship with symptoms, and the changes of these markers in the postoperative period will be evaluated.

DETAILED DESCRIPTION:
Serum Annexin V, sVCAM-1, sICAM-1, vascular endothelial growth factor and proinflammatory cytokines (TNF-a and interleukin-6) values were studied by taking blood samples from all patients before and three months after the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Stage III and IV endometriosis patients requiring surgery due to chronic pelvic pain or suspected malignancy

Exclusion Criteria:

1. Malignant disease
2. Ovarian failure
3. Acute pelvic inflammatory disease
4. Smokers
5. Pregnancy
6. Chronic autoimmune disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Stage III and IV endometriosis patients aged 18-50 years requiring surgery for chronic pelvic pain or suspected malignancy
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic value of serum Annexin V in endometriosis | Up to 4 months
  To determine whether serum Annexin V levels (ng/mL) can be used as diagnostic markers of endometriosis disease.
Diagnostic value of serum sVCAM-1 in endometriosis | Up to 4 months
  To determine whether serum sVCAM-1(ng/mL) levels can be used as diagnostic markers of endometriosis disease.
Diagnostic value of serum sICAM-1 in endometriosis | Up to 4 months
  To determine whether serum sICAM-1(ng/mL) levels can be used as diagnostic markers of endometriosis disease.
Diagnostic value of serum Vascular Endothelial Growth Factor in endometriosis | Up to 4 months
  To determine whether serum Vascular Endothelial Growth Factor (pg/mL) levels can be used as diagnostic markers of endometriosis disease.
Diagnostic value of serum TNF-alpha in endometriosis | Up to 4 months
  To determine whether serum TNF-alpha (pg/mL) levels can be used as diagnostic markers of endometriosis disease.
Diagnostic value of serum Interleukin-6 in endometriosis | Up to 4 months
  To determine whether serum Interleukin-6 (pg/mL) levels can be used as diagnostic markers of endometriosis disease.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Ebru Kovalak, MD, Principal Investigator — Bagcilar Training and Research Hospital
Locations (1):
- Bagcilar Teaching and Research Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vodolazkaia A, El-Aalamat Y, Popovic D, Mihalyi A, Bossuyt X, Kyama CM, Fassbender A, Bokor A, Schols D, Huskens D, Meuleman C, Peeraer K, Tomassetti C, Gevaert O, Waelkens E, Kasran A, De Moor B, D'Hooghe TM. Evaluation of a panel of 28 biomarkers for the non-invasive diagnosis of endometriosis. Hum Reprod. 2012 Sep;27(9):2698-711. doi: 10.1093/humrep/des234. Epub 2012 Jun 26. PMID 22736326
- See also: Based on the above publication — https://pubmed.ncbi.nlm.nih.gov/22736326/